CLINICAL TRIAL: NCT01662258
Title: Microbiology Testing With the Aim Of Directed Antimicrobial Therapy For Community-Acquired Pneumonia
Brief Title: Microbiology Testing With the Aim Of Directed Antimicrobial Therapy For CAP
Acronym: NIHCAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision by NIH
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Louisville (Other); Louisville VA Medical Center (U.S. Federal Agency); Johns Hopkins University (Other); Summa Health System (Other); Baylor College of Medicine (Other); Ben Taub Hospital (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HHSN272201000040C
Record Dates: First submitted 2012-08-03; First posted 2012-08-10 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Targeted strategy; Empiric therapy
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Point-of-Care diagnostic laboratory test (Experimental): Adult patients with community-acquired pneumonia (CAP) who are in the Targeted strategy group will undergo point-of-care (POC) diagnostic laboratory tests.
  Interventions: Device: Point-of-Care diagnostic laboratory test
- Empiric therapy (No Intervention): Option of no application of POC laboratory tests

INTERVENTIONS:
Device: Point-of-Care diagnostic laboratory test — All POC tests are FDA-cleared.
  Other Names: The POC tests are:; FilmArray (Idaho Tech, Salt Lake City, UT); Xpert Flu (Cepheid, Sunnyvale, CA); Vidas Brahms Procalcitonin (BioMerieux, Durham, NC); Urinary antigen for Strep pneumoniae (Alere, Waltham, MA); Legionella BinaxNOW urinary antigen(Alere, Waltham, MA); Gram stain of respiratory secretions
  Arms: Point-of-Care diagnostic laboratory test

SUMMARY:
This is a prospective interventional study to assess laboratory testing which will identify the microbial cause of pneumonia. This, in turn, will allow targeted antimicrobial agent selection for patients with community acquired-pneumonia (CAP).

Hypothesis: 1) To determine if Targeted strategy is non-inferior to Empiric therapy with respect to outcome endpoints. 2) To assess the use of innovative POC tests allows targeted narrow-spectrum antimicrobial therapy. 3) To determine if Targeted strategy is superior to Empiric therapy in patients with viral pneumonia

DETAILED DESCRIPTION:
The study will be conducted at five academic medical university sites with 7 hospitals. Empiric therapy is defined as selection of antibiotic therapy based on the 2007 ATS-IDSA guidelines in which broad-spectrum antibiotics are recommended, and microbial cause is uncertain

ELIGIBILITY:
Inclusion Criteria:

● Adult patients greater than age 17 years who are initially evaluated in the ED with symptoms of CAP. This includes those who will be treated as outpatients and those admitted to the hospital (both ward and ICU).

The definition of CAP is as follows:

* Presence of pulmonary infiltrates on chest radiography. (Initial reading may be performed by the ED physician - but has to be confirmed by board certified radiologist for inclusion in the study).
* At least 2 of the following: new onset of cough, productive sputum, shortness of breath, chest pain, fever > 380C, abnormal chest auscultation, WBC > 12,000 cells/mL.
* Able to provide informed consent
* Read, signed, and dated informed consent document
* Available for follow-up for the planned duration of the study

Exclusion Criteria:

* Patients with underlying immunosuppressive illness (HIV, neutropenia, asplenia, transplant recipient, cystic fibrosis, receipt of immunosuppressive medications including corticosteroids, (equivalent of prednisone > 10 mg) cancer chemotherapy, or anti-tumor necrosis factor agents.
* Patients residing in long-term care facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improvement or resolution of symptoms of CAP AND absence of objective signs of deterioration | 30 days after enrollment
  Symptoms of sputum, cough, shortness of breath. Objective signs of deterioration: Acute Respiratory Distress Syndrome, empyema,nonpulmonary infection by infecting microbe, ICU admission, rehospitalization within 7 days following discharge

SECONDARY OUTCOMES:
Identification of microbial etiology by laboratory testing | 30 days following enrollment, although microbial identification usually occurs within 5 days.
  POC microbiology testing including gram stain of respiratory secretions, blood culture, molecular probes.

OTHER OUTCOMES:
Receipt of narrow spectrum antimicrobial agent targeted toward a specific microbe (as opposed to empiric antimicrobial therapy that is broad-spectrum) | 30 days after enrollment although most patients will be evaluable within 5 days
  Antiviral agents will be administered at POC (point-of-care) if Influenza virus is identified by molecular testing. Penicillin compounds will be administered if Strep pneumoniae is identified. Macrolides/quinolone will be administered if Mycoplasma pneumoniae and Legionella are identified. Etc.
Length of stay (LOS) for hospitalized patients | 30 days after enrollment
  Educational measures using evidence-based endpoints for clinical response will lead to shorter LOS without concomitant increase in complications or clinical failure.

CONTACTS AND LOCATIONS:
Overall Officials: Victor L Yu, M.D., Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel, New York, New York
  - Summa Health System, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas